CLINICAL TRIAL: NCT00742820
Title: Randomized, Controlled, 3-Arm, Open Label, Cross-Over Bioequivalence Study Comparing Liquid PhosLo vs. PhosLo Gelcaps Using Calcium Citrate as a Positive Control in Healthy Volunteers
Brief Title: Bioequivalence Study Comparing Calcium Acetate Oral Solution Versus Calcium Acetate Gelcaps in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Fresenius Medical Care North America (Industry)
Responsible Party: Jonathan Greenberg, MD, Director Clinical Research, Fresenius USA Manufacturing Inc., d/b/a Fresenius Medical Care North America
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: LP-RTG-01-01
Record Dates: First submitted 2008-08-26; First posted 2008-08-28 (Estimated); Last update posted 2009-02-09 (Estimated); Status verified 2009-02

CONDITIONS: Hyperphosphatemia
Keywords: bioequivalence
MeSH Terms: conditions — Hyperphosphatemia | interventions — calcium acetate; Calcium Citrate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- 1 (Experimental): Calcium Acetate Oral Solution 667 mg per 5 mL
  Interventions: Drug: Calcium Acetate Oral Solution 667 mg per 5 mL
- 2 (Active Comparator): Calcium Acetate 667 mg Gelcaps
  Interventions: Drug: Calcium Acetate 667 mg GelCaps
- 3 (Other): Calcium Citrate 950 mg Caplets
  Interventions: Dietary Supplement: Calcium Citrate 950 mg Caplets

INTERVENTIONS:
Drug: Calcium Acetate Oral Solution 667 mg per 5 mL — Drug: Calcium acetate oral solution 667 mg calcium acetate, USP per 5 mL (169 mg of elemental calcium per 5 mL); Dosage: 30 mL of calcium acetate oral solution; Dosage frequency: three times per day with meals; Duration: 3 days and the morning of day 4, in total ten doses
  Arms: 1
Drug: Calcium Acetate 667 mg GelCaps — Drug: PhosLo GelCaps (calcium acetate) 667 mg (169 mg of elemental calcium per gelcap); Dosage: 6 gelcaps; Dosage frequency: three times per day with meals; Duration: 3 days and the morning of day 4, in total ten doses.
  Arms: 2
Dietary Supplement: Calcium Citrate 950 mg Caplets — Drug: Calcium Citrate 950 mg Caplets (200 mg of elemental calcium per caplet); Dosage: 5 caplets; Dosage frequency: three times per day with meals; Duration: 3 days and the morning of day 4, in total ten doses
  Arms: 3

SUMMARY:
To compare the bioequivalence of calcium acetate oral solution vs. calcium acetate gelcaps in healthy volunteers with calcium citrate as a positive control.

ELIGIBILITY:
Inclusion Criteria:

* Signed and dated informed consent form
* Ages: 18-75 years
* Serum Calcium level 8.6-10.2 mg/dL
* 25 vitamin D level 20-100 ng/mL
* 1, 25 dihydroxy vitamin D level 6-62 pg/mL
* Fasting glucose level of 65-99 mg/dL (min 8 hr fast)
* iPTH level of 10-65 pg/mL
* Serum phosphorous level of 2.5-4.5 mg/dL
* Albumin level of 3.6-5.1 g/dL
* Sodium level of 135-146 mEq/L
* Potassium level of 3.5-5.3 mEq/L
* Negative pregnancy test (at screening and prior to dosing) for women of childbearing potential and subjects must agree to use adequate contraception (hormonal or double barrier method) during the study
* No clinically significant abnormalities on electrocardiogram (ECG) reading as determined by the INVESTIGATOR
* No clinically significant abnormalities on liver function tests
* No clinically significant abnormalities on CBC and coagulation studies
* No clinically significant abnormalities on kidney function (eGFR using serum creatinine)
* BMI between 18.5-30
* Subjects must agree not to consume alcohol while in the treatment phase of the study

Exclusion Criteria:

* Women who are pregnant or breast feeding
* Malignancy except squamous cell carcinoma of the skin
* Documented current acute or chronic disease
* Positive for human immunodeficiency virus (HIV), hepatitis B or hepatitis C
* Myocardial infarction within 6 months of study Day 0
* Parathyroidectomy within 6 months of study Day 0
* Gastrointestinal disorder associated with impaired absorption of oral medications
* Inability to swallow tablets or tolerate calcium acetate oral solution
* Hormonal therapy (except for contraceptives), immunotherapy or corticoid therapy
* Concurrent antibiotic treatment
* Any concurrent investigational treatment within 30 days of screening
* Unable or unwilling to comply fully with the protocol
* Diuretic therapy such as Thiazides, Furosemide (INN) or frusemide (former BAN) within one month before screening
* Subjects taking over-the-counter (OTC) or prescribed phosphorous or calcium containing supplements
* Subjects testing positive for drugs of abuse

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 46 (Actual)
Dates: Start 2008-08; Primary Completion 2008-11 (Actual); Study Completion 2008-11 (Actual)

PRIMARY OUTCOMES:
Serum Phosphate | 24 hrs
Urinary Calcium | 24 hrs

SECONDARY OUTCOMES:
Serum Calcium | 24 hrs
Urinary Phosphate | 24 hrs
Serum insulin and glucose | 6 hrs

CONTACTS AND LOCATIONS:
Overall Officials: Antoinette A. Pragalos, MD, Principal Investigator — Community Research
Locations (1):
- Community Research, Cincinnati, Ohio, United States